CLINICAL TRIAL: NCT01888796
Title: Effect of Linagliptin Therapy on Myocardial Diastolic Function in Patients With Type 2 Diabetes Mellitus
Brief Title: Diastolic Dysfunction in Patients With Type 2 Diabetes Mellitus
Acronym: Diast Dysfkt
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: bad recruitment of suitable participants, just 8 patients in one year
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-025; 2012-003858-81 (EudraCT Number); EK 113/13 (Other: Ethics Committee University Hospital Aachen)
Record Dates: First submitted 2013-06-20; First posted 2013-06-28 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-02

CONDITIONS: Diabetes Mellitus Type 2 (T2DM); Left Ventricular Diastolic Dysfunction
Keywords: T2DM; diastolic dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Ventricular Dysfunction, Left | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linagliptin (Active Comparator): Linagliptin 5 mg (tablets) once daily for 6 month
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Placebo (tablets) once daily for 6 month
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Linagliptin
  Other Names: Trade name Trajenta® by Boehringer Ingelheim (BI) Pharma GmbH & Co KG, Biberach, Germany
  Arms: Linagliptin
Drug: placebo
  Arms: Placebo

SUMMARY:
Examination of the effect of Linagliptin versus placebo on diastolic function in patients with type 2 diabetes mellitus and diastolic dysfunction as assessed by transthoracic echocardiography.

Furthermore the effect on serum levels of NT-pro BNP as a biomarker of heart failure will be investigated.

DETAILED DESCRIPTION:
Treatment:

The Patients will receive Linagliptin 5 mg QD or placebo for a period of 6 months.

The echocardiography and 24h RR measurement will be performed at baseline and 6 months after initiation of the therapy.

The blood chemistry (Glucose, HbA1c, BNP) will be evaluated at baseline as well as 3 and 6 months after initiation of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus Type 2
2. Age > 50 years
3. HbA1c > 7%
4. Left ventricular diastolic dysfunction determined by echocardiography as average E/é ≥13 or average E/é≥8 and LA volume ≥34ml/m2
5. Stable anti-diabetic medication for the last 6 weeks which should include a maximal tolerated dose of metformin (unless contraindication or intolerance to metformin does exist).
6. Indication to increase anti-diabetic medication as judged by the investigator
7. Written informed consent prior to study participation

Exclusion Criteria:

1. Diabetes mellitus type 1
2. Echocardiography:

   * decreased left ventricular systolic function, ejection fraction (EF) <45%
   * regional wall motion abnormalities
   * hypertrophic cardiomyopathy (septum >15mm)
   * severe valvular dysfunction
3. Uncontrolled hypertension
4. Atrial fibrillation
5. Obstructive sleep apnea syndrome
6. Use of DPP-4 Inhibitor (Dipeptidyl-peptidase IV Inhibitor), GLP 1 agonists, Thiazolindinedione
7. Kidney disease CKD 4 and more (GFR < 30 ml/min/1.73)
8. Liver disease (ALT or AST > 3 times the upper limit of norm) or known liver cirrhosis
9. Active malignant disease
10. HbA1c > 8.5%
11. Recent (<3 months) clinically significant coronary or cerebral vascular event
12. Pregnant females as determined by positive [serum or urine] hCG test at Screening or prior to dosing. Participants of child-bearing age should use adequate contraception as defined in the study protocol.
13. Lactating females
14. The subject has a history of any other illness, which, in the opinion of the Investigator, might pose an unacceptable risk by administering study medication.
15. The subject received an investigational drug within 30 days prior to inclusion into this study
16. The subject has any current or past medical condition and/or required medication to treat a condition that could affect the evaluation of the study
17. The subject is unwilling or unable to follow the procedures outlined in the protocol
18. The subject is mentally or legally incapacitated

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular diastolic function | baseline and 6 months
  Change in left ventricular diastolic function between baseline and after 6 month as determined by 2D and novel 3D parameter global Strain Rate E Change in left ventricular diastolic function between baseline and after 6 month as determined by standardized parameter E/é and left atrial (LA) volume

SECONDARY OUTCOMES:
Change in serum NT-pro BNP levels | baseline and 6 months
  Change in serum NT-pro BNP levels

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, Univ.-Prof., Principal Investigator — Department of Internal Medicine I, RWTH Aachen University Hospital
Locations (1):
- Department of Internal Medicine I, University Hospital, Aachen, Germany